CLINICAL TRIAL: NCT00858455
Title: A Phase I, Open Label, Randomized, Four-Period Crossover Study to Evaluate the Effects of Maalox® Advanced Maximum Strength and One A Day® Maximum on Pharmacokinetics of GSK1349572 in Healthy Adult Subjects
Brief Title: A Study to Evaluate the Effect of Antacid and Multivitamin and Mineral Tablet on the Study Drug GSK1349572
Acronym: DDI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Shionogi (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 111602; ING111602
Record Dates: First submitted 2009-01-22; First posted 2009-03-09 (Estimated); Last update posted 2009-06-05 (Estimated); Status verified 2009-05

CONDITIONS: Healthy Volunteer
Keywords: Healthy Volunteers; Drug interation, Pharmacokinetics
MeSH Terms: interventions — dolutegravir

ARMS (1):
- Healthy Volunteers (Experimental): 4 period cross over
  Interventions: Drug: GSK1349572 and MaaloxAdvanced Maximum Strength; Drug: GSK1349572 and Maalox Advanced Maximum Strength; Drug: GSK1349572 and One A Day; Drug: GSK1349572

INTERVENTIONS:
Drug: GSK1349572 and MaaloxAdvanced Maximum Strength — A single dose of GSK1349572 co-administered with a single dose of 20 mL of Maalox Advanced Maximum Strength
Drug: GSK1349572 and Maalox Advanced Maximum Strength — A single dose of GSK1349572 administered 2 hours prior to administration of a single dose of 20 mL of Maalox Advanced Maximum Strength
Drug: GSK1349572 and One A Day — A single dose of GSK1349572 50 mg co-administered with a single dose of a One A Day Maximum multivitamin
Drug: GSK1349572 — A single dose of GSK1349572

SUMMARY:
The purpose is to study the effect of Maalox® and One A Day® on the pharmacokinetics of GSK1349572, and also to compare the safety of GSK1349572 when administered alone and when administered with Maalox® and One A Day®. There are four dosing periods in this study, each period requires a 4 night stay. A follow-up visit is also required at approximately 7 days after the last dose administration. Starting from the first period to the follow-up, it will take about 1 month. Screening visit is required to be completed within 30 days prior to the first dose.

MAALOX® is a registered trademark of Novartic Consumer Health, LLC. ONE A DAY® is a registered trademark of Bayer Healthcare LLC.

ELIGIBILITY:
Inclusion Criteria:

* A subject will be eligible for inclusion in this study only if all of the following criteria apply:
* Healthy as determined by a responsible physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* Male or female between 18 and 65 years of age.
* A female subject is eligible to participate if she is of non-childbearing potential (i.e., physiologically incapable of becoming pregnant) including any female who:
* Is pre-menopausal with a documented bilateral tubal ligation, bilateral oophorectomy (removal of the ovaries) or hysterectomy, or
* Is post-menopausal defined as 12 months of spontaneous amenorrhea. A follicle stimulating hormone (FSH) level will be performed to confirm a postmenopausal status. For this study, FSH levels > 40 mlU/ml is confirmatory. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt, HRT should be discontinued for 2 weeks and then the subject rescreened, as HRT can suppress FSH.
* Male subjects must agree to use one of the contraception methods listed in Section 8.1. This criterion must be followed from the time of the first dose of study medication until 14 days after the last dose of study medication.
* Body weight ≥ 50 kg for men and ≥ 45 kg for women and body mass index (BMI) within the range 18.5-31.0 kg/m2 (inclusive).
* AST, ALT, alkaline phosphatase and bilirubin ≤ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%). One repeat measurement to confirm eligibility is allowed.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* A subject will not be eligible for inclusion in this study if any of the following criteria apply:
* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* History of sensitivity to any of the study medications, or components thereof, or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* If heparin is used during PK sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >14 drinks/week for men or >7 drinks/week for women. One drink is equivalent to (12 g alcohol) = 5 ounces (150 ml) of wine or 12 ounces (360 ml) of beer or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication.
* Pregnant females as determined by positive serum or urine human chorionic gonadotrophin (hCG) test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Subjects with a history of cholecystectomy should be excluded.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive Hepatitis B surface antigen or positive Hepatitis C antibody result.
* A positive test for HIV antibody.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject's systolic blood pressure is outside the range of 90-140mmHg, or diastolic blood pressure is outside the range of 45-90mmHg or heart rate is outside the range of 50-100bpm for female subjects or 45-100 bpm for male subjects. A single repeat to determine eligibility is allowed.
* Exclusion criteria for screening ECG as specified in the protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Single dose plasma GSK1349572 PK parameters including AUC(0-∞), Cmax, and C24 will be obtained to compare single dose plasma GSK1349572 PK with that of GSK1349572 after dministration with Maalox and One A Day as per the study design in the protocol | PK samples will be commected and analyzed starting with pre-dose and going for up to 72 hours post dose in each period in each study period

SECONDARY OUTCOMES:
Safety and tolerability parameters, including adverse event, concurrent medication,clinical laboratory, ECG, and vital signs assessments. Single dose plasma GSK1349572 PK parameters: AUC(0-t), AUC(0-24), tlag, tmax, CL/F, and t1/2. | Data will be collected from Dosing until the final follow-up after completion of all study periods.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Buffalo, New York, United States